CLINICAL TRIAL: NCT01179659
Title: A Pharmacokinetic Study to Assess the Bioequivalence of a Single-Dose of KUDCO and Wyeth Pharmaceuticals (Protonix) 40 mg Pantoprazole Sodium Delayed-Release Tablet When Administered to Healthy Adult Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of Pantoprazole 40 mg DR Tablets and Protonix 40 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kremers Urban Development Company (Industry)
Responsible Party: Gartano Morelli, MD, MDS Pharma Services
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP872
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Single dose crossover BE study
MeSH Terms: interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protonix (Active Comparator): Protonix 40 mg DR Tablet (Wyeth Pharmaceuticals)
  Interventions: Drug: Pantoprazole 40 mg DR Tablet vs. Protonix 40 mg DR Tablet
- Pantoprazole 40 mg DR Tablet (Experimental): Pantoprazole 40 mg DR Tablet vs. Protonix 40 mg DR Tablet
  Interventions: Drug: Pantoprazole 40 mg DR Tablet vs. Protonix 40 mg DR Tablet

INTERVENTIONS:
Drug: Pantoprazole 40 mg DR Tablet vs. Protonix 40 mg DR Tablet — Single dose crossover BE study

SUMMARY:
The objective of this study was to assess the single-dose bioequivalence of KUDCO's and Wyeth Pharmaceuticals' (Protonix) 40 mg pantoprazole sodium delayed-lease tablets, under fed conditions.

DETAILED DESCRIPTION:
This was an open-label, randomized, fully replicated crossover, 2-sequence bioequivalence study under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, non-smoking (for at least 6 months) male or female volunteers, 18 - 55 years of age.
* Weighed at least 52 kg for males and 45 kg for females and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983).
* Medically healthy subjects with clinically normal laboratory profiles, vital signs, and ECG.
* Females of childbearing potential were either sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study, or using one of the following acceptable birth control methods:

  1. Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum.
  2. Intrauterine device (IUD) in place for at least 3 months.
  3. Barrier method (condom, diaphragm) with spermicide for at least 14 days prior to the first dose and throughout the study.
  4. Surgical sterilization of the partner (vasectomy for 6 months minimum).
  5. Hormonal contraceptives for at least 3 months prior to the first dose of the study.
* Gave voluntary written informed consent to participate in the study.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
* In addition, history or presence of:

  1. Alcoholism or drug abuse within the past 2 years;
  2. Hypersensitivity or idiosyncratic reaction to pantoprazole, omeprazole, or any other substituted benzimidazole proton-pump. inhibitors.
* Females who were pregnant or lactating.
* History of tobacco use or use of products containing nicotine (i.e., smoking cessation aids such as nicotine gum or patches) within the 6 months prior to the first dose.
* Subjects who tested positive at screening for human immunodeficiency virus (HIV) antibody screen, hepatitis B surface antigen screen (HbsAg), or hepatitis C antibody screen (HCV).
* Treatment with any known enzyme-altering drugs (barbiturates, phenothiazines, cimetidine, etc.) within 30 days prior to the first dose.
* Difficulty in swallowing medication or any gastrointestinal disease that would affect the drug absorption.
* Subjects who had been on a special diet (for whatever reason) during the 28 days prior to the first dose and throughout the study.
* Subjects who, through completion of the study, would have donated in excess of:

  * 500 mL of blood in 14 days;
  * 1500 mL of blood in 180 days;
  * 2500 mL of blood in one years.
* Subjects who participated in another clinical trial with 28 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2005-09; Primary Completion 2005-11 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum observed concentration of drug substance in plasma) | 26 hours
AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration) | 26 hours
AUC0-inf (area under the concentration-time curve from time zero to infinity) | 26 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano morelli, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Saint-Laurent, Montreal, Quebec, Canada